CLINICAL TRIAL: NCT05941052
Title: Supporting, Mobilizing and Accelerating Research for Tuberculosis Elimination (SMART4TB)- Technical Area (TA) 1: Diagnostics- Assessing Diagnostics At Point-of-care for Tuberculosis (ADAPT)
Brief Title: Assessing Diagnostics At Point-of-care for Tuberculosis
Acronym: ADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University Hospital Heidelberg (Other); KNCV Tuberculosis Foundation (Other); Bingham University (Unknown); University of California, Irvine (Other); De La Salle University Medical Center (Other); Centre for Infectious Disease Research in Zambia (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7200AA22RFA00004
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Diagnostics; Global Health
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Evaluation of various novel TB triage and diagnostic tests (Experimental): For the novel TB triage and diagnostic tests, the investigators will conduct large-scale evaluation of design-locked tests in a cohort of adults with presumed TB. The investigators aim to enroll 450 participants per year at each of three enrollment sites for evaluation of various novel TB triage and diagnostic tests and 50 health workers to assess test usability.
  Interventions: Diagnostic Test: Tongue swab-based molecular assays

INTERVENTIONS:
Diagnostic Test: Tongue swab-based molecular assays — The investigators will evaluate semi-automated or automated molecular assays intended for use at near point of care or point of care.

SUMMARY:
Every year, more than 3 million people with TB remain undiagnosed and 1 million die. Better diagnostics are essential to reducing the enormous burden of TB worldwide. The Assessing Diagnostics At Point-of-care for Tuberculosis (ADAPT) study seeks to reduce the burden of TB worldwide by evaluating faster, simpler, and less expensive TB triage and diagnostic tests.

DETAILED DESCRIPTION:
The Assessing Diagnostics At Point-of-care for Tuberculosis (ADAPT) seeks to identify and rigorously assess promising, design-locked point-of-care (POC) tuberculosis (TB) diagnostic tests (hereafter referred to as "novel tests") in clinical studies conducted in settings of intended use. Rapid diagnosis and effective treatment are critical for improving patient outcomes and reducing TB transmission. However, nearly one-third of people with TB are not diagnosed or reported to public health authorities.The different types of tests required to reduce this "diagnostic gap" have been described in the form of target product profiles (TPPs) defined by the World Health Organization (WHO). The highest priority TPP is that for a point-of-care, non-sputum biomarker-based test to facilitate rapid TB diagnosis using easily accessible samples (i.e., a biomarker-based diagnostic test). The ADAPT study will evaluate the sensitivity, specificity and yield of novel diagnostic tests against a reference standard including sputum Xpert® Mycobacterium tuberculosis/Rifampicin (MTB/RIF) Ultra and sputum mycobacterial culture among adolescents and adults with presumptive TB (based on having TB symptoms, or TB risk factor + positive TB screening test) presenting to outpatient health facilities in high burden countries. In addition, the usability and acceptability of novel TB diagnostic tests will be assessed through direct observations and surveys of routine health workers.

ELIGIBILITY:
Novel TB triage and diagnostic tests:

Inclusion Criteria-

The investigators will include non-hospitalized adults (age ≥ 12 years) with either:

1. cough ≥2 weeks' duration, a commonly accepted criterion for identifying people with presumed pulmonary TB (to facilitate standardization across sites and comparison of test performance across sub-groups; OR
2. risk factors for which TB screening is recommended (HIV infection, self-reported close contact, history of mining work). People with risk factors will be included if they screen positive for TB based on WHO-recommended screening tools as specified below:

Positive TB screening definitions by risk factor:

1. People Living with Human Immunodeficiency Virus (PLHIV) (Risk Factor): C Reactive Protein (CRP) >5 mg/dL OR abnormal chest x-ray (CXR)
2. Self-reported Close Contact (Risk Factor): abnormal CXR History of mining work (Risk Factor): abnormal CXR

Exclusion Criteria-

1. Completed latent or active TB treatment within the past 12 months (to increase TB prevalence and reduce false-positive results, respectively);
2. Have taken any medication with anti-mycobacterial activity (including fluoroquinolones) for any reason, within 2 weeks of study entry (to reduce false-negatives);
3. Reside >20km from the study site or are unwilling to return for follow-up visits; OR
4. Are unwilling to provide informed consent

Assessment of the usability of novel TB tests:

Inclusion Criteria-

The investigators will include health workers at each clinical site who are:

1. aged ≥18 years; AND
2. involved in routine TB testing (collecting specimens for or performing TB tests).

Exclusion Criteria-

The investigators will exclude staff who are:

1) unwilling to provide informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion with positive index test result among participants with tuberculosis (TB) | 2 years
  Sensitivity - Number with positive index test result/(Number with positive or negative index t test result) among participants with TB. TB will be defined based on a microbiological reference standard (sputum mycobacterial culture results)
Proportion with negative index test result among participants without tuberculosis (TB) | 2 years
  Specificity - Number with negative index test results/(Number with positive or negative index t test result) among participants without TB. TB will be defined based on a microbiological reference standard (sputum mycobacterial culture results)

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Cattamanchi, Principal Investigator — University of California, Irvine
Locations (3):
- Zankli Research Center, Bingham University, Abuja, Nigeria
- De La Salle Medical and Health Sciences Institute, Dasmariñas, Philippines
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SN, Brennan PJ. Tuberculosis: diagnostics. Tuberculosis (Edinb). 2007 Aug;87 Suppl 1:S14-7. doi: 10.1016/j.tube.2007.05.001. Epub 2007 Jun 20. PMID 17584529
- [Background] World Health Organization. Global tuberculosis report Geneva, Switzerland: World Health Organization, 2015.
- [Background] Organization WH. High-priority target product profiles for new tuberculosis diagnostics: report of a consensus meeting. Geneva, Switzerland: WHO Press, 2014.
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Walusimbi S, Bwanga F, De Costa A, Haile M, Joloba M, Hoffner S. Meta-analysis to compare the accuracy of GeneXpert, MODS and the WHO 2007 algorithm for diagnosis of smear-negative pulmonary tuberculosis. BMC Infect Dis. 2013 Oct 30;13:507. doi: 10.1186/1471-2334-13-507. PMID 24172543
- [Background] Xpert MTB/RIF Implementation Manual: Technical and Operational 'How-To'; Practical Considerations. Geneva: World Health Organization; 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK254323/ PMID 25473699
- [Background] Subbaraman R, Nathavitharana RR, Satyanarayana S, Pai M, Thomas BE, Chadha VK, Rade K, Swaminathan S, Mayer KH. The Tuberculosis Cascade of Care in India's Public Sector: A Systematic Review and Meta-analysis. PLoS Med. 2016 Oct 25;13(10):e1002149. doi: 10.1371/journal.pmed.1002149. eCollection 2016 Oct. PMID 27780217